CLINICAL TRIAL: NCT01402336
Title: 'A Multicentre, Prospective Randomized Study to Assess the Effect When GnRH Antagonist is Started Either on Stimulation Day 1 and Day 6 vs. Conventional GnRH Agonist Long Protocol in Patients With Polycystic Ovary Syndrome Undergoing IVF-ET
Brief Title: GnRH Antagonist Versus GnRH Agonist in Polycystic Ovary Syndrome During in Vitro Fertilization - Embryo Transfer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Young Min Choi, Young Min Choi, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCOS_IVF
Record Dates: First submitted 2011-07-04; First posted 2011-07-26 (Estimated); Last update posted 2017-10-10 (Actual); Status verified 2017-10

CONDITIONS: Infertility; Polycystic Ovary Syndrome
Keywords: Polycystic ovary syndrome; ovulation induction; In vitro fertilization-embryo transfer
MeSH Terms: conditions — Infertility; Polycystic Ovary Syndrome | interventions — cetrorelix; Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- GnRH antagonist, SD #1 starting group (Experimental): Start GnRH antagonist from stimulation day 1 during ovulation induction cycles
  Interventions: Drug: GnRH antagonist (Cetrorelix)
- GnRH antagonist, SD #6 starting group (Experimental): Start GnRH antagonist from stimulation day 6 during ovulation induction cycles
  Interventions: Drug: GnRH antagonist (Cetrorelix)
- Conventional GnRH agonist long group (Active Comparator): Conventional GnRH agonist long protocol
  Interventions: Drug: Conventional GnRH agonist (Triptorelin)

INTERVENTIONS:
Drug: GnRH antagonist (Cetrorelix) — In the first arm, cetrotide will be administrated from the first day during stimulation. In the second arm, cetrotide will be administrated from the sixth day during stimulation
  Other Names: Cetrotide
  Arms: GnRH antagonist, SD #1 starting group; GnRH antagonist, SD #6 starting group
Drug: Conventional GnRH agonist (Triptorelin) — Patients in the agonist group were administered GnRH agonist started 5 days before discontinuation of the oral contraceptive.
  Other Names: Decapeptyl
  Arms: Conventional GnRH agonist long group

SUMMARY:
GnRH (Gonadotropin-releasing hormone) antagonists in IVF (in vitro fertilization) has been accomplished by several randomized controlled trials compared with conventional GnRH agonist long protocol in polycystic ovary syndrome (PCOS) patients. Moreover, there are debating issues that refer to the timing of GnRH antagonist initiation. The purpose of this study is to investigate the laboratory and clinical priority during ovarian stimulation for IVF in patients with PCOS treated with three different protocols.

DETAILED DESCRIPTION:
GnRH Antagonist is Started on Stimulation Day 1 GnRH Antagonist is Started on Stimulation Day 6 Conventional GnRH Agonist Long Protocol

ELIGIBILITY:
Inclusion Criteria:

* PCOS patients (diagnosed as 2003 ASRM(The American Society for Reproductive Medicine)/ESHRE(The European Society of Human Reproduction and Embryology) consensus meeting guideline)
* age 20-40 years
* patients who have normal uterus
* Korean ethnicity

Exclusion Criteria:

* patients who have abnormal thyroid function
* patients who have abnormal prolactin test
* patients who have diabetes, or Cushing's syndrome, or congenital adrenal hyperplasia, or androgen-producing tumor.
* Patients who reject informed consent
* patients who have experience of adverse events for GnRH agonist, antagonist, recombinant FSH(follicle-stimulating hormone).

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2011-06; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
number of oocyte retrieved | ovum pick up day, At the point of ovum pick-up, we can count how many oocyte was retrieved. So, almost just after ovum pick-up, outcome measure will be possible.

SECONDARY OUTCOMES:
pregnancy rate | after confirming fetal heart beat via transvaginal ultrasound. Usually 2~4 weeks after ovum pick-up day.

CONTACTS AND LOCATIONS:
Overall Officials: Young Min Choi, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea